CLINICAL TRIAL: NCT01848574
Title: Satisfaction Understanding of Patients and Relatives in Emergency Room
Acronym: SUPER4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NI10067
Record Dates: First submitted 2013-02-19; First posted 2013-05-07 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: All Inpatient in Short Stays Emergencies
Keywords: Understanding; Patients; Emergency; Information
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual procedure (No Intervention): Investigators will give medical information to their patients as usual.
- Experimental procedure (Experimental): You must use the standardized patient information. The final Information of the patient before the final output should be clear and concise in the presence of trustworthy people if the patient wishes.
  Deliver the following information in the orde of the items below:
  Decline your identity and function Provide a final diagnosis, indicating the affected organ and Inform prognosis (any severity), and the potential duration of affection
  Briefly additional tests:
  * Radio show
  * Explain the main abnormalities Explain treatment modalities and setpoint monitoring Finish with an open question: "Do you have questions? "If you think the state anxiety or depression alters the patient's understanding, still deliver all the information listed above.
  Interventions: Other: standardized multifaceted information procedure to improve patients' comprehension

INTERVENTIONS:
Other: standardized multifaceted information procedure to improve patients' comprehension
  Arms: Experimental procedure

SUMMARY:
Evaluation of global understanding and with items of patients admitted to the emergency.

Prospective observational study randomized in cluster during 6 weeks in 14 centers

DETAILED DESCRIPTION:
Patients' comprehension in the emergency department (ED) is relatively low. This is more evident for in-patients with more complex diseases. The preliminary study conducted suggests that patients' comprehension was improved by the use of standardized information and by opening a dialogue. This study however had its limits. It does not deliver proper information guideline to physicians working in the ED.

This study is reproduced on a larger scale for in-patients in the ED concerning their comprehension about the medical information given and thus improving the scientific evidence. This study has been conducted on a national level in 2 phases with 14 investigating centers spread in Paris and other provinces:

First, an observational period was conducted during 2 weeks in each center in order to document their homogeneity. At the same time, this period permitted to have a reference level of comprehension. During this period, investigators continued to give medical information to their patients as usual. The aim is to adjust the results of the comprehensions levels in 2 groups after the experimental study on the "baseline" data.

Second, an experimental period of 4 weeks: 7 centers are identified as "formal procedure group" and their investigators are provided with formal procedures on the patient's comprehension in the ED based on updated literature data. At the same time, recommendations are given on the information given to patients. 7 other centers "control group" only formal presentation on the patient's comprehension in the ED on updated literature data.

According to the center where the patient is included, he will be either in the "formal procedure group" or the "control group".

Among all in-patients in the ED, it is planned to include:

* 700 patients in the observational period (50 in each center)
* 1400 patients in the experimental period (700 in the formal procedure group and 700 in the control group)

Improvement in the information given to patients is expected due to the participation of the centers in this study. This improvement is expected in both arms only due to the fact of their participation. Better information level is expected in the "formal procedure group".

If this study proves a better information in the procedure group, then our aim will be to propose recommendations to ED physicians to improve the information given to in-patients in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over
* Inpatient Unit in Short Term Hospitalization (UHCD)
* Patient who agreed to participate in the study
* Patient affiliated to a social security scheme (beneficiary or righ)

Exclusion Criteria:

* Patient has already been included in the study, which was re-hospitalized for the same reason UHCD
* Patient in judicial restraint (certificate of non-admission in custody, incarcerated)
* Patient for which a decision forced hospitalization was taken
* Patient non-Francophone
* Patients with underlying cognitive and unable to give their consent
* Patient opposed to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1816 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Global Comprehension | Day 0
  Completing the questionnaire independently by the doctor and the patient after patient and physician interview final and comparison of responses

SECONDARY OUTCOMES:
Comprehension of each items | Day 0
  Completing the questionnaire independently by the doctor and the patient after patient and physician interview final and comparison of responses

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Erick Claessens, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France